CLINICAL TRIAL: NCT06156111
Title: Bacterial Microleakage and Bone Loss in Internal Connection Dental Implants Based on the Type of Abutment Used in Zirconia Partial Fixed Prosthesis: in Vivo Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Principal Investigator, Miguel Gómez Polo, Associate Professor of Conservative Dentistry and Prosthodontics, Universidad Complutense de Madrid
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18/426-E
Record Dates: First submitted 2023-11-20; First posted 2023-12-05 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Jaw, Edentulous, Partially
Keywords: Dental implants; Dental abutments; Dental prosthesis; Dental implant-abutment; Implant-Abutment Connections
MeSH Terms: conditions — Jaw, Edentulous, Partially | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Prospective double-blinded, randomized, paired sample (split-mouth).
Who Masked: Participant, Investigator
Masking Description: The assessment and the measurements will be performed by a separate person, not the operator. The patient will not know in which quadrant the abutments will be placed or not.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transepithelial abutment (Other): The patients randomized to the transepithelial abutment group will receive a fixed screw implant-supported zirconia prosthesis which will be attached to the implants through an implant-abutment connection.
  Interventions: Device: Transepithelial abutment group
- Direct to implant (Experimental): The patients randomized to the direct to implant group will receive a fixed screw implant-supported zirconia prosthesis which will be attached direct to the implants connection.
  Interventions: Device: Direct to implant group

INTERVENTIONS:
Device: Transepithelial abutment group — Before completing the essential clinical data registration to produce an individual patient-oriented prosthesis, trans-epithelial abutments on the implants randomized to this group will be put at the torque the manufacturer recommends (30 Ncm typically), according to the appropriate gingival height and then the fixed implant-supported monolithic zirconia will be placed at the torque of 15 Ncm
  Other Names: Control Group
  Arms: Transepithelial abutment
Device: Direct to implant group — It will be registered the essential clinical data registration to produce an individual patient-oriented prosthesis, and then the fixed implant-supported monolithic zirconia will be placed at the torque of 30 Ncm.
  Other Names: Test Group
  Arms: Direct to implant

SUMMARY:
This clinical trial aims to observe if there are differences in bacterial micro-filtration on interfaces and to evaluate if there are differences in the occurrence of peri-implant diseases and bone loss in fixed partial monolithic zirconia CAD/CAM implantsupported prostheses with and without abutment in patients at the Advanced Implant Prosthetics Clinic of the Complutense University of Madrid, of both sexes, over 18 years of age, whose treatment plan is based on the replacement of dental pieces with two fixed partial dentures on implants, in such a way that the study will be performed "split mouth" rehabilitating one of them with zirconia bridges on attachments with connection and others with Zirconia bridges with flat attachments or without connection. The main question it aims to answer is whether the not use of abutment influence bacterial micro-leakage and the development of peri-implant diseases and bone loss at that level in fixed partial monolithic zirconia CAD/CAM prothesis.

Participants will:

* Receive two fixed partial monolithic zirconia CAD/CAM prothesis, one will be attached to an abutment (control group) and the other not (test group)
* Subsequently, control appointments of the fixed implant supported prosthesis treatment will be performed (1, 3,6, 12 and 24 months) and radiographies will be made with the parallelizing device attached by the silicone key.

Researchers will compare fixed partial monolithic zirconia CAD/CAM implant-supported prostheses with and without abutment to see:

* Differences in bacterial micro-leakage on interfaces.
* Occurrence of peri-implant diseases and bone loss

DETAILED DESCRIPTION:
BACKGROUND

Since the discovery of osseointegration by Branemark, dental implant treatment has been growing in importance for the replacement of missing teeth until it has become the treatment of choice in most cases of partial and total tooth absences. Although in the beginning, implants were used to hold mandibular prostheses, they had a smooth surface, and the connection they presented on their platform was an external hexagon. These characteristics were established empirically in the absence of previous experience. Currently, implants are one of the most widely used dental treatments and have evolved both in their indications and in their design. Regarding their indications, they are used for the treatment of all types of edentulism, from a unitary implant to the rehabilitation of a complete arch. On the other hand, in terms of design, the modifications and variables are so numerous that it is impossible to list them all, but fundamentally, it has progressed on the surface, macroscopically and microscopically, achieving a greater proportion of tooth-implant union, and in the connection, moving from the initial external hexagon to internal connections with different designs: hexagonal, octagonal, morse cone, and hexagon, with the aim of preventing the complications that can appear in this type of prosthesis, both mechanical (the most frequent being loosening of the screw) and biological (mainly bacterial microfiltration).

The mismatch at the level of the junction between implant-abutment or implant-prosthesis in the case of a prosthesis directly screwed to the implant(s) has been and is one of the workhorses in implantology due to the influence it has on bacterial microfiltration, and this is demonstrated by the large number of studies that exist on this subject. In an ideal situation, this mismatch should not exist and should be cero, so that the bacteria existing in the oral microflora could not filter and accumulate in that implant attachment or implant prosthesis junction. In reality, it is impossible to achieve that perfection goal even in the manufacture of prefabricated machined parts and for unit implants, since a dimensional margin is necessary to allow their correct settlement, especially when connected directly to the implant (without the intermediation of a prefabricated abutment) by individualized manufacturing processes. That is why, from this point of view, it would be advisable to use prefabricated abutments in all cases of partial prostheses in order to keep the possible misalignment of the prosthesis away from the implant-attachment joint. This mismatch, however, must be understood not only as evaluated by different studies as a linear discrepancy but also from a three-dimensional point of view, since once it is accepted that the perfect fit does not exist, microfiltration will occur to a greater or lesser extent depending on the design of the connection; for example, it will not be the same in an external hexagonal connection as in an internal octagonal one.

The importance of bacterial microfiltration at the level of the implant-abutment junction from a clinical point of view is of special relevance since the accumulation of bacteria at that level, in most cases subgingival, could be directly related to the colonization of anaerobic bacteria, more aggressive, in locations that are difficult to access for sanitization by the patient. in such a way that they could favor the beginning of pathological bone destruction and the development of a peri-implant disease, complications of relative frequency, and that can be defined as infectious processes that occur in the tissues around the implants. When the inflammation around the implants presents with bone loss, bleeding, and/or suppuration on probing, it is considered peri-implantitis. It is a complication that is complicated and difficult to treat since the surface of the implant is contaminated and non-surgical treatments are usually insufficient to clean it, while surgical treatments are not only more aggressive but are also not inflatable and can also lead to aesthetic complications due to retraction of the soft tissues and even the exposure of the implant itself (metallic in most cases).

On the other hand, as for the implant prosthesis itself, its evolution since its origins with respect to its design and materials has also been very important. Among the materials used today to make fixed prostheses on implants, one of the most important is zirconia. Its use has become widespread because it has qualities that improve the materials considered until recently the gold standard, which were made with a metal structure (Titanium, Cr-Co, Cr-Ni, Cr-Ni, Cr-Ni-Pa, Pa-Co, etc.) and the aesthetic coating of porcelain, added by a brushstroke process carried out by a laboratory technician and then fired in processing ovens. Among the advantages of zirconia are: its CAD/CAM (Computer Aided Design/Computer Aided Manufacturing) manufacturing, i.e., computer design and manufacturing by milling process (as it can be milled in a softer, pre-synthesized phase, improves metal milling, makes it cheaper, and involves much less wear); its biocompatibility; and its aesthetics, as it is a white material. This quality allows the creation of prostheses without the need for aesthetic coating, known as monolithic zirconium. This modality, monolithic zirconium, is one of the most used treatment alternatives in fixed prostheses on implants because it also manages to solve one of the most frequent mechanical complications in fixed prostheses on implants, which is the porcelain jump or chipping. The term "chipping" is defined as "the detachment of one material attached to another when subjected to a load, separating the two".

When prostheses are rehabilitated on teeth with monolithic zirconia, the procedure is similar to the gold standard (metal-porcelain); however, when rehabilitating prostheses on implants, we must consider that the peculiarities of zirconia discourage its direct screwing to the implant since its lower resistance to compressive forces in thin thicknesses causes them to fracture at the moment of definitive tightening of the prosthesis (torques of 30-40 Ncm). In addition, in the event of loosening of the prosthesis, its great hardness means that the movements between the implant and prosthesis cause the internal surface of the connection to be worn, which can even lead to the need to remove the implant as it becomes unusable. For this reason, monolithic zirconium on implants is made on metal abutments or interfaces, to which it is joined by a cementing process. Within these attachments, when used in implants with internal connection, there are those with connection (they fit into the implant connection) or flat or without connection (they remain at the level of the implant platform but do not penetrate it). The latter are easier to use in all cases since the implant-abutment fit is easier and hardly complicated in cases of angled implants, but they leave an "unfilled" space within the internal surface of the implant, which could lead to greater bacterial microfiltration, with the possible influence on the development of peri-implant diseases that has been explained above.

Based on this background, the following in vivo study is carried out to assess whether the use of connected or unconnected abutments influences bacterial microfiltration, the development of peri-implant diseases, and bone loss at that level in partial prostheses on monolithic zirconia CAD/CAM implants.

HYPOTESIS

Taking into account the importance of microfiltration at the level of the implant-abutment junction and its relationship with the development of peri-implant diseases, and the increase in fixed implant rehabilitations performed by CAD/CAM in monolithic zirconia, its study is considered of great importance, proposing the following hypotheses and objectives:

* Null hypothesis 1: There are no differences in bacterial microfiltration in partial prostheses performed by CAD/CAM in monolithic zirconium with abutments and without abutments.
* Null hypothesis 2: there are no differences in the development of peri-implant diseases and bone loss in partial prostheses performed using CAD/CAM in monolithic zirconium with abutments and without abutments.

OBJECTIVES

1. To observe if there are differences in bacterial microfiltration in fixed partial implant-supported prostheses performed by CAD/CAM in monolithic zirconium with and without abutment.
2. Assess whether there are differences in the occurrence of peri-implant diseases and bone loss in partial prostheses performed by CAD/CAM in monolithic zirconium with abutment and without abutment.

These objectives are in line with those proposed by the State Research Agency in its call for R+D+i research projects "RESEARCH CHALLENGES", being identified within the challenge "Health, demographic change, and well-being", being considered relevant within oral prosthetic treatments, and also being highly topical objectives whose contribution, with the aim of being published in journals within the Journal of Citation Report, will have an impact on the treatment of implant prostheses and their incidence in the development of peri-implantitis and peri-implant diseases.

MATERIAL AND METHODS

Study design

Longitudinal parallel prospective double blinded clinical trial.

Study population

The study population will consist of patients seen at the School of Dentistry of the Complutense University of Madrid, of both sexes, over 18 years of age, who require as treatment the replacement of teeth with two fixed partial prostheses supported by implants and who meet all the inclusion criteria but none of the exclusion criteria. This way the study could be carried out "with a split mouth" design rehabilitating one of them with zirconia bridges with abutments connection and others with zirconia bridges with unconnected abutments.

Once the informed consent has been read and explained, and any possible doubts regarding the treatment and the study have been resolved, patients must give their written informed consent to participate in the study prior to any study-related procedure.

Study Sample and sample size

15 patients will be selected who come for treatment at the school of Dentistry of Complutense University of Madrid and who require as treatment the replacement of teeth with two fixed partial prostheses on implants, in such a way that the study will be carried out "with a split mouth".

Methodology: Clinical procedures, data colection and information sources

Patients will be given the patient information sheet and will be explained any questions that may arise, as well as informed consent. The patient may revoke his or her participation in the study at any time he or she deems appropriate and without the need to give explanations.

Implants will be placed where there is sufficient bone availability and at least 4 months have elapsed since the only extraction, excluding locations where there are infectious focus or where bone regeneration procedures have been needed.

The prosthetic phase will be shifted following the osseointegration period. Prior to that, a parallelization technique will be used to take an initialx-ray. A silicone key will be made to help reposition the parallelizer in the same position so that all subsequent X-rays will be obtained in the same perspective, allowing for the monitoring of bone resorption, if it occurs.

In order to submit the models to the laboratory for the creation of the monolithic zirconia bridges-one on the implant-abutment connection and the other on the implant-crown connection-the appropriate records will need to be taken. Randomization will be used to determine which bridge will have abutments.

The fixed implant-supported prosthesis will undergo control/follow-up appointments at the first month and then every 3, 6, 12, and 24 months. During each appointment, peri-apical X-rays will be taken using the parallelizing device, which is held in place by the silicone key.

Ultimately, the images will be exported to a computer program (Image J/Photoshop) in which the radiographic loss will be measured for each follow-up period.

It will be verified during the patient's follow-up that there have been no biological or mechanical issues.The implants will be probed to assess bleeding at probing (BOP), document the presence of plaque, and study the peri-implant tissues to ascertain if they are healthy or have mucositis or peri-implantitis.

Additionally, a microbiological examination will be conducted, involving the collection of a sample using paper tips from the adjacent teeth and the implant conection of all implants in both study groups. The samples will then undergo PCR analysis to detect the presence of periodontopathogenic bacteria. Only patients who have had their restorations placed on implants and had at least a year of follow-up will have this microbiological sample obtained.

In the same methodical manner as when the prosthesis was placed, the occlusion and contact points will be examined, and their thickness will be measured using thickness sheets. Furthermore, an intraoral scan using the 3Shape Trios scanner will be carried out in order to assess any volumetric changes generated at the soft tissue level and determine whether the restorations or antagonists have worn down.

A questionnaire will be carried out, evaluating patient satisfaction (Annex 2d.).

STATISTICAL ANALYSIS

Since there are fewer than twenty samples in each group (n < 20), the Kolmogorov-Smirnov will be used to determine whether the samples meet normal criteria. The ANOVA test for independent samples will be used in this study to statistically assess the fracture resistance as well as the level of microfiltration, provided that the normality criteria are met. All the examining variables are quantitative and independent. The non-parametric Kruskal-Wallis test for independent samples will be used instead if this condition is not satisfied.

STUDUY LIMITATIONS

The study's main limitations is the recruitment of patients since they have to be patients with edentations that allow their treatment with both types of prostheses for controlled comparison, that is, split mouth. In addition, they must be in good health and have good bone availability, which makes them susceptible to inclusion in the study.

CHRONOGRAM / WORK PLAN

Since the approval of the research project:

* Year 1: Detailed review of the new bibliography, fabrication of the in vitro study samples, and beginning of methodology (estimated: application of cyclic loading and 1/2 thermocycling in all groups). Patient selection, in vivo study, and implant placement
* Year 2: Continuation with the thermocycling phase and completion of the in vitro phase (bacterial infiltration and obtaining results), continuing with patient selection and implant placement, and beginning of the prosthetic phases of the implants already placed.
* Year 3: In vitro study: obtaining results, statistical analysis, and writing them for publication in JCR journals; clinical phase: continuation of case selection, alternating placement of implants (if cases are still missing),

PROTOCOL AMENDMENTS Protocol changes will be kept to a minimum. Only those changes that are deemed essential to the successful completion of the protocol will be considered.

PUBLICATION RIGHTS

Analysis of data will be conducted by Data Management. The final manuscript will be prepared by the principal investigator in conjunction with sub-investigators and submitted for publication. Additionally, the results of the study will be entered on clinicaltrials.gov.

If it's decided on the future sharing of the IPD the following data will be shared and available:

* Participant's data that underlie the results reported in this article, after identification (text, tables, figures).
* The data and protocols may be only available to investigators and researchers who provide a methodologically sound proposal for individual participant data meta-analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients susceptible to treatment with implants.
* Being over 18 years old.
* Not being severe smokers (>20 cigarettes/day)
* Not having diseases that can affect bone metabolism, such as arthritis and osteoporosis, and not having uncontrolled systemic diseases.

Exclusion Criteria:

* Any contraindications for oral surgical procedures.
* Conditions or circumstances that, in the opinion of the investigator, would preclude completion of participation in the study or interfere with the analysis of the study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-02-26 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Bacterial micro-filtration: Bacterial load analysis | 2 years
  Samples will be obtained at the conection of the study control and study test from each patient. Samples will be taken with two consecutive sterile medium paper-points (#30, Maillefer, Ballaigues, Switzerland) that were kept in place for 30 s and then transferred into a screw-capped vial. Samples will be transported to the microbiology laboratory within 2 h and stored in deep freezing (-80ºC). Samples will be processed for multiplex RTPCR for detection of total anaerobic counts and counts of selected periodontal pathogens Data will be expressed in colony-forming units (CFU) per mL of the original sample.
Bone level change | 2 years
  On the standardized peri-apical radiographs implant bone levels will be evaluated. The reference point for the bone level measurement will be the implant shoulder. The bone level will be measured as the distance between the implant shoulder and the first visible bone contact on the implant. Mean bone level changes between two time-points will be computed by subtracting the average bone level from one visit with the other.
Peri-implant pathologies development | 2 years
  The peri-implant pathologies development will be evaluated through the presence of unhealthy clinical records on probing pocket depth and bleeding on probing.

SECONDARY OUTCOMES:
Probing pocket depth (PPD) | 2 years
  The PPD will be measured around the implant by recording the distance in millimeters from the gingival margin to the bottom of the pocket at 6 locations (meso-vestibular, disto-vestibular, vestibular, meso-palatal, palatal/lingual, disto-palatal).
Bleeding on Probing (BoP) | 2 years
  Bleeding on probing (BoP) will be recorded according to Lang et al. 1986. The presence or absence of bleeding on probing (BoP) will be documented as a "yes" or "no" on 6 sites (meso-vestibular, disto-vestibular, vestibular, meso-palatal, palatal/lingual, disto-palatal).
Inter-proximal contact point | 2 years
  Inter-proximal contact point will be evaluated in millimeters (mm) using an inter proximal contact gauge for a precise inter-proximal measurement.
Prosthetic mechanical behavior | 2 years
  The prosthetic mechanical behavior will be evaluated through prosthetic survival/success based on the occurrence of some mechanical complications. The mechanical complications to be evaluated will be classified by visual inspection in clinical examination as follows:
  * Appearance of material skips, minor fractures and/or chipping, loosening of occlusal screw
  * Appearance of major fractures defined as an appearance of a broken structure that restrain the use of the protheses.
Patient satisfaction | 2 years
  The Spanish version of the abbreviations OHIP-14 and OHIP-49, will be utilized in this study. The original OHIP-49 is the source of the OHIP-14. OHIP-49 is Functional limitation, physical pain, psychological discomfort, physical disability, psychological disability, social impairment, and handicap are the seven domains that make up its 49 items. The OHIP-14, which has 14 items across these seven areas, has shown to be responsive to modifications in oral health and prosthetic therapy. Subjects are asked how often they have experienced each occurrence over the past month for each question. On a Lickert scale, responses are scored as follows: 0 = never, 1 = seldom, 2 = occasionally, 3 = frequently, 4 = very frequently, and 5 = constantly. A low OHRQoL is indicated by a high OHIP score (41).
Protheses material wear | 2 years
  An intraoral scanner (Trios, 3Shape) was used to measure in millimeters (mm) the protheses material wear at different timepoints. Using a 3D computer software (Geomagic) the STLs from all the scans of each protheses were superimposed to evaluate the three-dimensional soft tissue changes during follow-up.
Volumetric variation of peri-implant soft tissues | 2 years
  An intraoral scanner (Trios, 3Shape) was used to measure in millimeters (mm) the soft tissue changes different timepoints. Using a 3D computer software (Geomagic) the STLs from all the scans of each protheses were superimposed to evaluate the three-dimensional soft tissue changes during follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Gómez Polo, DDS, PhD, Principal Investigator — UComplutense de Madrid
Locations (1):
- School of Dentistry, Complutense University. Pza Ramón y Cajal s/n., Madrid, Spain

REFERENCES:
- [Background] Smith NA, Turkyilmaz I. Evaluation of the sealing capability of implants to titanium and zirconia abutments against Porphyromonas gingivalis, Prevotella intermedia, and Fusobacterium nucleatum under different screw torque values. J Prosthet Dent. 2014 Sep;112(3):561-7. doi: 10.1016/j.prosdent.2013.11.010. Epub 2014 Mar 20. PMID 24656409
- [Background] Baldassarri M, Hjerppe J, Romeo D, Fickl S, Thompson VP, Stappert CF. Marginal accuracy of three implant-ceramic abutment configurations. Int J Oral Maxillofac Implants. 2012 May-Jun;27(3):537-43. PMID 22616046
- [Background] Larrucea C, Conrado A, Olivares D, Padilla C, Barrera A, Lobos O. Bacterial microleakage at the abutment-implant interface, in vitro study. Clin Implant Dent Relat Res. 2018 Jun;20(3):360-367. doi: 10.1111/cid.12589. Epub 2018 Feb 15. PMID 29446238
- [Background] Alves DCC, de Carvalho PSP, Elias CN, Vedovatto E, Martinez EF. In vitro analysis of the microbiological sealing of tapered implants after mechanical cycling. Clin Oral Investig. 2016 Dec;20(9):2437-2445. doi: 10.1007/s00784-016-1744-0. Epub 2016 Feb 20. PMID 26895757
- [Background] Elshiyab SH, Nawafleh N, George R. Survival and testing parameters of zirconia-based crowns under cyclic loading in an aqueous environment: A systematic review. J Investig Clin Dent. 2017 Nov;8(4). doi: 10.1111/jicd.12261. Epub 2017 Mar 19. PMID 28317331
- [Background] Gehrke SA, Delgado-Ruiz RA, Prados Frutos JC, Prados-Privado M, Dedavid BA, Granero Marin JM, Calvo Guirado JL. Misfit of Three Different Implant-Abutment Connections Before and After Cyclic Load Application: An In Vitro Study. Int J Oral Maxillofac Implants. 2017 Jul/Aug;32(4):822-829. doi: 10.11607/jomi.5629. PMID 28708914
- [Background] Bressan E, Stocchero M, Jimbo R, Rosati C, Fanti E, Tomasi C, Lops D. Microbial Leakage at Morse Taper Conometric Prosthetic Connection: An In Vitro Investigation. Implant Dent. 2017 Oct;26(5):756-761. doi: 10.1097/ID.0000000000000657. PMID 28945671
- [Background] Guerra E, Pereira C, Faria R, Jorge AO, Bottino MA, de Melo RM. The Impact of Conical and Nonconical Abutments on Bacterial Infiltration at the Implant-Abutment Interface. Int J Periodontics Restorative Dent. 2016 Nov/Dec;36(6):825-831. doi: 10.11607/prd.2779. PMID 27740643
- [Background] Butignon LE, Basilio Mde A, Pereira Rde P, Arioli Filho JN. Influence of three types of abutments on preload values before and after cyclic loading with structural analysis by scanning electron microscopy. Int J Oral Maxillofac Implants. 2013 May-Jun;28(3):e161-70. doi: 10.11607/jomi.2481. PMID 23748335
- [Background] Butignon LE, de Almeida Basilio M, Santo JS, Arioli Filho JN. Vertical Misfit of Single-Implant Abutments Made from Different Materials Under Cyclic Loading. Int J Oral Maxillofac Implants. 2016 Sep-Oct;31(5):1017-22. doi: 10.11607/jomi.4477. PMID 27632255
- [Background] Larrucea Verdugo C, Jaramillo Nunez G, Acevedo Avila A, Larrucea San Martin C. Microleakage of the prosthetic abutment/implant interface with internal and external connection: in vitro study. Clin Oral Implants Res. 2014 Sep;25(9):1078-83. doi: 10.1111/clr.12217. Epub 2013 Jul 4. PMID 23822097
- [Background] Colpani JT, Borba M, Della Bona A. Evaluation of marginal and internal fit of ceramic crown copings. Dent Mater. 2013 Feb;29(2):174-80. doi: 10.1016/j.dental.2012.10.012. Epub 2012 Dec 4. PMID 23218747
- [Background] Kim KB, Kim JH, Kim WC, Kim JH. Three-dimensional evaluation of gaps associated with fixed dental prostheses fabricated with new technologies. J Prosthet Dent. 2014 Dec;112(6):1432-6. doi: 10.1016/j.prosdent.2014.07.002. Epub 2014 Sep 11. PMID 25218032
- [Background] Fernandez M, Delgado L, Molmeneu M, Garcia D, Rodriguez D. Analysis of the misfit of dental implant-supported prostheses made with three manufacturing processes. J Prosthet Dent. 2014 Feb;111(2):116-23. doi: 10.1016/j.prosdent.2013.09.006. Epub 2013 Oct 28. PMID 24176182
- [Background] Tartaglia GM, Sidoti E, Sforza C. Seven-year prospective clinical study on zirconia-based single crowns and fixed dental prostheses. Clin Oral Investig. 2015 Jun;19(5):1137-45. doi: 10.1007/s00784-014-1330-2. Epub 2014 Oct 12. PMID 25304166
- [Background] Guess PC, Att W, Strub JR. Zirconia in fixed implant prosthodontics. Clin Implant Dent Relat Res. 2012 Oct;14(5):633-45. doi: 10.1111/j.1708-8208.2010.00317.x. Epub 2010 Dec 22. PMID 21176095
- [Background] Lang NP, Berglundh T; Working Group 4 of Seventh European Workshop on Periodontology. Periimplant diseases: where are we now?--Consensus of the Seventh European Workshop on Periodontology. J Clin Periodontol. 2011 Mar;38 Suppl 11:178-81. doi: 10.1111/j.1600-051X.2010.01674.x. PMID 21323713
- [Background] Zarone F, Russo S, Sorrentino R. From porcelain-fused-to-metal to zirconia: clinical and experimental considerations. Dent Mater. 2011 Jan;27(1):83-96. doi: 10.1016/j.dental.2010.10.024. Epub 2010 Nov 21. PMID 21094996